CLINICAL TRIAL: NCT01308684
Title: Open-label, Combined Dose-finding (Phase I) and Efficacy-finding (Phase II) Study of RO5323441 in Combination With Bevacizumab for Patients With Recurrent Glioblastoma
Brief Title: A Dose- and Efficacy-Finding Study of RO5323441 in Combination With Avastin (Bevacizumab) in Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP25389; 2010-021795-29
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — TB-403; Bevacizumab

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RO5323441 + bevacizumab [Avastin]
- 2 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]

INTERVENTIONS:
Drug: RO5323441 + bevacizumab [Avastin] — Dose-Finding part: RO5323441 intravenous escalating doses once every two weeks; Efficacy-Finding part: established dose from the Dose-Finding part; Avastin: 10 mg/kg intravenously once every two weeks
  Arms: 1
Drug: bevacizumab [Avastin] — Efficacy-Finding part: 10 mg/kg intravenously once every two weeks
  Arms: 2

SUMMARY:
This open-label, multicenter study will evaluate the safety and efficacy of RO5323441 in combination with Avastin (bevacizumab) in patients with recurrent glioblastoma. In the dose-finding part, patients will receive intravenous escalating doses of RO5323441 in combination with 10 mg/kg Avastin once every two weeks. In the efficacy-finding part, patients will be randomized to receive the established dose (from the dose-finding part) of RO5323441 plus Avastin or Avastin alone. Patients in the dose-finding part may continue treatment with RO5323441 and Avastin on the study until evidence of progressive disease or unacceptable adverse events happen. In the efficacy-finding part, patients will receive study treatment until disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Histologically confirmed glioblastoma
* Radiographic demonstration of disease progression by Response Assessment in Neurooncology (RANO) criteria following prior therapy
* Availability of at least 1 formalin-fixed paraffin-embedded tumor tissue sample
* If receiving corticosteroids, patients must have been on a stable or decreasing dose of corticosteroids
* Prior standard radiotherapy for glioblastoma
* Karnofsky Performance status >/=70
* Over 4 weeks since prior surgical resection
* Over 12 weeks from radiotherapy
* Over 4 weeks from anticancer agents

Exclusion Criteria:

* Patients had second or later glioblastoma relapse
* Patients received more than one systemic treatment regimen for glioblastoma
* Patients have secondary glioblastoma
* Prior treatment with Avastin
* Patients unable to undergo Magnetic Resonance Imaging (MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Dose-Finding Part: Dose limiting toxicity | Day 28
Efficacy-Finding part: Progression-free survival | From baseline to disease progression or death (>12 months)

SECONDARY OUTCOMES:
Dose-Finding part: Pharmacokinetics of RO5323441 and Avastin when combined | From baseline to disease progression or death (>12 months)
Dose-Finding part: Safety (incidence of adverse events) | From baseline to disease progression or death (>12 months)
Dose-Finding part: Efficacy (tumor response according to Response Assessment in Neurooncology (RANO) criteria | From baseline to disease progression or death (>12 months)
Dose-Finding part: Glioblastoma biomarker | From baseline to disease progression or death (>12 months)
Efficacy-Finding part: Overall Response Rate | From baseline to disease progression or death (>12 months)
Efficacy-Finding part: Disease Control Rate | From baseline to disease progression or death (>12 months)
Efficacy-Finding part: Duration of Response | From baseline to disease progression or death (>12 months)
Efficacy-Finding part: Progression-free survival | From baseline to disease progression or death (>12 months)
Efficacy-Finding part: Overall Survival | From baseline to disease progression or death (>12 months)
Efficacy-Finding part: Safety (incidence of adverse events) | From baseline to disease progression or death (>12 months)
Efficacy-Finding part: Glioblastoma biomarker | From baseline to disease progression or death (>12 months)
Efficacy-Finding part: Pharmacokinetics (serum levels) of RO5323441 and Avastin when combined | From baseline to disease progression or death (>12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- København Ø, Denmark
- Marseille, France
- Zurich, Switzerland
- Manchester, United Kingdom